CLINICAL TRIAL: NCT03400683
Title: Different Methods of Termination of Second Trimester Abortion: Comparative Clinical Study
Brief Title: Different Methods of Termination of Second Trimester Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Induction of Abortion
MeSH Terms: interventions — Misoprostol; Letrozole; Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- misoprostol only group (Active Comparator): given 200 microgram misoprostol (Misotac 200 microgram tablet, Sigma Pharmaceuticals, Egypt), in sublingual every four hours for a maximum of five doses
  Interventions: Drug: Misoprostol
- misoprostol with letrozole group (Active Comparator): group received 15mg( letrozole2.5mg) on three successive day patient take doses of letrozole for daily oral three successive day at home by herself and forth day admitted to our hospital followed by sublingual misoprostol 200 microgram misoprostol (Misotac 200 microgram tablet, Sigma Pharmaceuticals, Egypt), every four hours for a maximum of five doses
  Interventions: Drug: Misoprostol; Drug: Letrozole
- misoprotol with Foley's catheter group (Active Comparator): the transcervical 16F Foley's catheter with 30 ml balloon capacity (Euromed for Medical Industries, Cairo, Egypt, under license of Kanglite, USA), inserted under aseptic conditions withsublingual misoprostol 200 microgram misoprostol (Misotac 200 microgram tablet, Sigma Pharmaceuticals, Egypt), every four hours for a maximum of five doses
  Interventions: Drug: Misoprostol; Procedure: Foley's catheter

INTERVENTIONS:
Drug: Misoprostol — 200 microgram misoprostol in sublingual every four hours for a maximum of five doses
  Other Names: Misotac
Drug: Letrozole — 15mg( letrozole 2.5mg) on three successive day
  Other Names: Femara
  Arms: misoprostol with letrozole group
Procedure: Foley's catheter — transcervical 16F Foley's catheter with 30 ml balloon capacity inserted under aseptic conditions
  Other Names: Urinary catheter
  Arms: misoprotol with Foley's catheter group

SUMMARY:
The Patient are divided into 3 groups group 1 included 50 cases using misoprostol only. group 2 included also 50 cases in which using misoprostol with letrozole. Group3 included also 50 cases in which using misoprostol with Foleys catheter for termination of second trimesteric abortion between 14 and 24 weeks

DETAILED DESCRIPTION:
Pregnant women were randomized into three equal groups: Group allocation was blindly randomized concealed by placement in numbered opaque sealed envelopes. These envelopes were kept in the labor ward and drawn in consecutive order:

Group 'A" (misoprostol only group): Pharmacological method for termination of second trimester missed abortion was done by given 200 microgram misoprostol (Misotac 200 microgram tablet, Sigma Pharmaceuticals, Egypt), in sublingual every four hours for a maximum of five doses.

Group 'B'(misoprostol with letrozole group): The anti-estrogen action of letrozole has been show to be useful in pretreatment for termination of pregnancy ,in combination with misoprostol,women in the letrozole group received 15mg( letrozole2.5mg) on three successive day patient take doses of letrozole for daily oral three successive day at home by herself and forth day admitted to our hospital followed by sublingual misoprostol 200 microgram misoprostol (Misotac 200 microgram tablet, Sigma Pharmaceuticals, Egypt), every four hours for a maximum of five doses.

Group 'C' (misoprotol with Foley's catheter group): Mechanical method for termination of second trimester missed abortion was done using the transcervical 16F Foley's catheter with 30 ml balloon capacity (Euromed for Medical Industries, Cairo, Egypt, under license of Kanglite, USA), inserted under aseptic conditions withsublingual misoprostol 200 microgram misoprostol (Misotac 200 microgram tablet, Sigma Pharmaceuticals, Egypt), every four hours for a maximum of five doses.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* gestational age between 14 and 24 weeks
* Fetal death was confirmed by ultrasonic scan
* Unfavorable cervix using Bishop score for cervical assessment with score less than 5
* Parity less than 5
* No uterine contractions

Exclusion Criteria:

* Previous uterine scar eg scar for cessarian section
* Rupture of membranes
* Chorioamnionitis
* Placenta previa or low lying placenta.
* Women with medical disease like DM, coagulopathy or genital infections.
* Hypersensitivity or contraindications for receiving misoprostol, including:Maternal asthma.Sickle cell disease.Known hypersensitivity to prostaglandins.History of glaucoma

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
complete evacuation of uterus | 24 hours after treatment
  clear endometrial line < 4 mm in thickness

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided